CLINICAL TRIAL: NCT01683565
Title: Preemie Tots: A Pilot Study to Understand the Effects of Prematurity in Toddlerhood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sarah Keim (Other)
Collaborators: Cures Within Reach (Other); Marci and Bill Ingram Fund for Autism Spectrum Disorders Research (Unknown)
Responsible Party: Sponsor-Investigator, Sarah Keim, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 752311
Record Dates: First submitted 2012-09-04; First posted 2012-09-12 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Preterm Birth; Child Development; Child Behavior
MeSH Terms: conditions — Premature Birth; Child Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCPUFA Oil Supplement (Experimental): EPA + DHA + GLA + OA oil supplement
  Interventions: Drug: LCPUFA oil supplement
- Canola Oil Placebo (Placebo Comparator)
  Interventions: Other: Canola Oil Placebo

INTERVENTIONS:
Drug: LCPUFA oil supplement — 2.5mL per day for 90 days
  Daily Dose: EPA (338mg) + DHA (225mg) + GLA (83mg) + OA (200mg)
  Arms: LCPUFA Oil Supplement
Other: Canola Oil Placebo — 2.5mL per day for 90 days
  Arms: Canola Oil Placebo

SUMMARY:
The purpose of this study is to examine whether supplementation with certain polyunsaturated fatty acids can help development and behavior of children born preterm.

ELIGIBILITY:
Inclusion Criteria:

1. Child born at less than or equal to 29 completed weeks' gestation;
2. Child between 18 months, 0 days and 38 months, 30 days old chronological age;
3. Child admitted to NICU and/or had a Neonatology Clinic follow up visit scheduled.
4. Child showing some autistic symptoms;
5. Child between the 5th and 95th percentiles (per WHO growth chart) for weight at his/her most recent hospital visit;
6. English spoken in the home, demonstrate ability to communicate in English well-enough to understand study, informed consent, and study questionnaires; and
7. Have informed consent on file.

Exclusion Criteria:

1. Consume LCPUFA supplement drops, chews, powders, Pediasure, or fatty fish more than 2x per week;
2. Unable to tolerate venipuncture;
3. Any major malformation that would preclude participation;
4. Cerebral Palsy (quadriparesis only);
5. Deafness;
6. Blindness;
7. Bleeding disorder;
8. Type I diabetes;
9. Fragile X Syndrome, Rett Syndrome, Angelman Syndrome, Tuberous Sclerosis;
10. Non febrile seizure in the last month without a clear and resolved etiology;
11. Feeding problem that may inhibit full participation;
12. Known fish allergy;
13. Known canola/rapeseed allergy or sensitivity; or
14. Recorded score of <70 on Bayley Cognitive Section within the past year.

Ages: 18 Months to 39 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Keim, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Boone KM, Klebanoff MA, Rogers LK, Rausch J, Coury DL, Keim SA. Effects of Omega-3-6-9 fatty acid supplementation on behavior and sleep in preterm toddlers with autism symptomatology: Secondary analysis of a randomized clinical trial. Early Hum Dev. 2022 Jun;169:105588. doi: 10.1016/j.earlhumdev.2022.105588. Epub 2022 May 19. PMID 35644107
- [Derived] Keim SA, Gracious B, Boone KM, Klebanoff MA, Rogers LK, Rausch J, Coury DL, Sheppard KW, Husk J, Rhoda DA. omega-3 and omega-6 Fatty Acid Supplementation May Reduce Autism Symptoms Based on Parent Report in Preterm Toddlers. J Nutr. 2018 Feb 1;148(2):227-235. doi: 10.1093/jn/nxx047. PMID 29490101
- [Derived] Boone KM, Gracious B, Klebanoff MA, Rogers LK, Rausch J, Coury DL, Keim SA. Omega-3 and -6 fatty acid supplementation and sensory processing in toddlers with ASD symptomology born preterm: A randomized controlled trial. Early Hum Dev. 2017 Dec;115:64-70. doi: 10.1016/j.earlhumdev.2017.09.015. Epub 2017 Sep 20. PMID 28941976

RESULTS

PARTICIPANT FLOW:
Groups:
- Long Chain Polyunsaturated Fatty Acid (LCPUFA) Oil Supplement: Eicosapentaenoic acid (EPA) + Docosahexaenoic acid (DHA)
  + Gamma-Linolenic acid (GLA) + Oleic Acid (OA)
  LCPUFA oil supplement: 2.5mL per day for 90 days
  Daily Dose: EPA (338mg) + DHA (225mg) + GLA (83mg) + OA (200mg
Period: Overall Study
Arm/Group | Long Chain Polyunsaturated Fatty Acid (LCPUFA) Oil Supplement | Canola Oil Placebo
Started | 15 | 16
Completed | 12 | 15
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Discontinued Intervention | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Long Chain Polyunsaturated Fatty Acid (LCPUFA) Oil Supplement | Canola Oil Placebo | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 16 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 30 [25 to 36] | 25 [23 to 25] | 27 [23 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 8 | 13 | 21
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Child Behavior - Pervasive Developmental Disorders Screening Test-II Stage 2
Description: The Pervasive Developmental Disorders Screening Test-II stage 2 (PDDST-II) is a 14-item measure designed to discriminate Autism Spectrum Disorders from a related non-autistic developmental disorder in children ages 12 to 48 months old. The min score is 0 and the max score is 14. Scores equal to or greater than five yield a positive screen for autism. PDDST-II scores were measured at baseline and then again at study completion (90 days post randomization). The scores were calculated as the PDDST-II value at 90 days minus the PDDST-II value at baseline.
Time Frame: Baseline to 90 days post randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long Chain Polyunsaturated Fatty Acid (LCPUFA) Oil Supplement | Canola Oil Placebo
Number analyzed (Participants) | 15 | 16
score on a scale | -1.0 (2.6) | -0.2 (1.9)
Statistical Analysis 1: Comparison: Long Chain Polyunsaturated Fatty Acid (LCPUFA) Oil Supplement vs Canola Oil Placebo; The sample size was determined based on the goal of confirming trial feasibility and estimating effect sizes for a full-scale trial, not for a definitive test of efficacy. The enrollment goal was 40, which would have provided an indication of an expected effect size for a larger full-scale trial (e.g., 53% power to detect a 2-point decrease (approximately 0.7-SD based on a prior study) in Pervasive Developmental Disorders Screening Test-II score). Funding limitations capped enrollment at 31; Test type: Other — Analyses compared the change in Pervasive Developmental Disorders Screening Test-II scores between groups, controlling for baseline scores, using mixed effects regression. This method leverages maximum likelihood to account for missing data. Treatment-by-time interaction terms were included as fixed effects and served as estimates of treatment effect. Group mean differences divided by the standard deviation were also calculated as effect sizes; p = 0.67, Mixed Models Analysis — Threshold for statistical significance (<0.05)

2. Primary Outcome: Child Behavior-Brief Infant-Toddler Social and Emotional Assessment (BITSEA)
Description: Brief Infant-Toddler Social and Emotional Assessment (BITSEA) is a 42 item tool that is useful for identifying social-emotional problems and/or deficits in children. BITSEA includes the following subscales: Competence (11 Items, min score:0, max score:22), problem behaviors--dysregulation (8 items, min score:0, max score:16) , externalizing (6 items, min score:0, max score:12), internalizing (8 items, min score:0, max score:16), Autism Spectrum Disorder (17 Items, min score:0, max score:34), and Red Flags (14 items, min score:0, max score:28).The questions overlap and the problem subscale is a combination of dysregulation, externalizing, and internalizing. Higher problem scores indicate greater levels of social-emotional/behavioral problems. Lower Competence scores indicate possible delay/deficit. Scores were measured at baseline and then again at study completion (90 days post randomization). The change in BITSEA scores were calculated as the value at 90 days - the value at baseline.
Time Frame: Baseline to 90 days post randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Long Chain Polyunsaturated Fatty Acids (LCPUFA) Supplement: Eicosapentaenoic acid (EPA) + Docosahexaenoic acid (DHA)
  + Gamma-Linolenic acid (GLA) + Oleic Acid (OA)
  LCPUFA oil supplement: 2.5mL per day for 90 days
  Daily Dose: EPA (338mg) + DHA (225mg) + GLA (83mg) + OA (200mg)
Arm/Group | Long Chain Polyunsaturated Fatty Acids (LCPUFA) Supplement | Canola Oil Placebo
Number analyzed (Participants) | 15 | 16
score on a scale
  Competence | 1.9 (3.2) | 0.9 (3.6)
  Problems | 3.2 (6.1) | -3.2 (5.0)
  Dysregulation | -0.9 (2.3) | -0.8 (2.2)
  Externalizing | 0.3 (1.3) | -0.7 (2.3)
  Internalizing | -0.9 (2.3) | -0.5 (2.3)
  Austism Spectrum Disorder | -1.5 (2.6) | 0.8 (3.8)
  Red Flag | -2.5 (3.8) | -1.0 (2.8)
Statistical Analysis 1: Comparison: Long Chain Polyunsaturated Fatty Acids (LCPUFA) Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in Competence scores between groups (LCPUFA vs. Placebo); Test type: Other — Analyses compared the change in BITSEA outcome scores between groups, controlling for baseline scores, using mixed effects regression. This method leverages maximum likelihood to account for missing data. Treatment-by-time interaction terms were included as fixed effects and served as estimates of treatment effect; no participant characteristics were included as covariates in the models. Group mean differences divided by the standard deviation were also calculated as effect sizes; p = 0.22, Mixed Models Analysis — Threshold for statistical significance (<0.05)
Statistical Analysis 2: Comparison: Long Chain Polyunsaturated Fatty Acids (LCPUFA) Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in Problem scores between groups (LCPUFA vs. Placebo); Test type: Other — Analyses compared the change in the BITSEA outcome scores between groups, controlling for baseline scores, using mixed effects regression. This method leverages maximum likelihood to account for missing data. Treatment-by-time interaction terms were included as fixed effects and served as estimates of treatment effect; no participant characteristics were included as covariates in the models. Group mean differences divided by the standard deviation were also calculated as effect sizes; p = 0.92, Mixed Models Analysis — Threshold for statistical significance (<0.05)
Statistical Analysis 3: Comparison: Long Chain Polyunsaturated Fatty Acids (LCPUFA) Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in Dysregulation scores between groups (LCPUFA vs. Placebo); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.88, Mixed Models Analysis
Statistical Analysis 4: Comparison: Long Chain Polyunsaturated Fatty Acids (LCPUFA) Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in Externalizing scores between groups (LCPUFA vs. Placebo); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.23, Mixed Models Analysis
Statistical Analysis 5: Comparison: Long Chain Polyunsaturated Fatty Acids (LCPUFA) Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in Internalizing scores between groups (LCPUFA vs. Placebo); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.91, Mixed Models Analysis
Statistical Analysis 6: Comparison: Long Chain Polyunsaturated Fatty Acids (LCPUFA) Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in Austism Spectrum Disorder scores between groups (LCPUFA vs. Placebo); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.03, Mixed Models Analysis
Statistical Analysis 7: Comparison: Long Chain Polyunsaturated Fatty Acids (LCPUFA) Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in Red Flag scores between groups (LCPUFA vs. Placebo); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.07, Mixed Models Analysis

3. Secondary Outcome: Fatty Acid
Description: The secondary outcome measures in this trial involve an examination of change in fatty acids from the first study visit to the final study visit.
Time Frame: Baseline to 90 days post randomization
Population: Rows titles are fatty acids with different C:D ratio where, "C" stands for Carbohydrate; "D" stands for Double bond; "C:D" is the ratio of the total amount of Carbon atoms of the fatty acid in relation to the number of double (unsaturated) bonds in it.
Measure: Mean (Standard Deviation); unit: nmol/mL
Groups:
- LCPUFA Oil Supplement: EPA + DHA + GLA + OA oil supplement
  LCPUFA oil supplement: 2.5mL per day for 90 days
  Daily Dose: EPA (338mg) + DHA (225mg) + GLA (83mg) + OA (200mg)
Arm/Group | LCPUFA Oil Supplement | Canola Oil Placebo
Number analyzed (Participants) | 13 | 15
nmol/mL
  10:0 | 2.15 (3.23) | -4.91 (7.37)
  12:0 | 2.56 (2.90) | -2.43 (6.68)
  14:0 | -3.07 (4.62) | -8.42 (6.84)
  16:0 | 177 (99.60) | -28.0 (116.05)
  16:1n-7 | 7.83 (9.90) | 27.0 (17.75)
  18:0 | 138 (69.25) | -40.3 (99.18)
  18:1n-9 | 80.5 (46.66) | -21.6 (50.19)
  18:1n-7 | 11.0 (4.98) | -2.13 (6.23)
  18:2n-6 | 18.7 (69.83) | -8.72 (56.53)
  18:3n-6 | 1.69 (2.54) | -4.29 (5.36)
  18:3n-3 | 2.44 (2.19) | -3.81 (5.50)
  18:4n-3 | -0.15 (1.19) | -3.44 (3.75)
  20:3n-6 | 6.24 (9.05) | -17.1 (15.30)
  20:4n-6 | 60.3 (57.74) | -7.72 (70.23)
  20:5n-3 | 38.7 (8.21) | -2.73 (12.90)
  22:5n-3 | -3.27 (4.88) | -2.84 (4.97)
  22:6n-3 | 109 (26.50) | -1.44 (26.69)
  total omega-6 | 86.9 (122.71) | -37.9 (138.07)
  total omega-3 | 146 (34.13) | -14.3 (43.64)
Statistical Analysis 1: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (10:0 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.31, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 2: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (12:0 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.47, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 3: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (14:0 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.38, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 4: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (16:0 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.02, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 5: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (16:1n-7 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.16, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 6: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (18:0 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.02, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 7: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (18:1n-9 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.02, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 8: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (18:2n-6 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.21, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 9: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (18:3n-6 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.34, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 10: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (18:3n-3 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.24, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 11: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (18:4n-3 nmol/mL ) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.50, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 12: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (20:3n-6 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.07, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 13: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (20:4n-6 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.10, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 14: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (20:5n-3 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.001, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 15: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (22:5n-3 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.71, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 16: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (22:6n-3 nmol/mL) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.001, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 17: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (Total Omega-6) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.10, t-test, 2 sided — P-values <0.05 were considered statistically significant
Statistical Analysis 18: Comparison: LCPUFA Oil Supplement vs Canola Oil Placebo; The reported p-value is for the comparison of the change in erythrocyte fatty acid composition (total omega-3) between groups (LCPUFA vs. Placebo); Test type: Other — Differences in mean changes in erythrocyte fatty acid composition were examined using t-tests; p = 0.10, t-test, 2 sided — P-values <0.05 were considered statistically significant

4. Other Pre Specified Outcome: Feasibility: Future Full-scale Multi-site Study
Description: Feasibility of a future full-scale multi-site study is assessed by examining the number of children screened, the proportion of these children who screen positive for ASD, the number of children who agree to participate in the trial, the number of children who return for the second and third study visits, baseline differences in individual fatty acids between the intervention and comparison groups, and adherence to the assigned treatment.
Time Frame: Pre-baseline to 90 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | LCPUFA Oil Supplement | Canola Oil Placebo
Number analyzed (Participants) | 15 | 16
Participants | 15 | 16

ADVERSE EVENTS:
Time Frame: Baseline to 90 days post randomization
Description: Information to be collected includes event description, time of onset, Study Doctor's assessment of severity, relationship to study product,and time of resolution/stabilization of the event. All AEs occurring during study participation must be documented appropriately regardless of relationship.
Arm/Group | LCPUFA Oil Supplement | Canola Oil Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 15/15 | 16/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCPUFA Oil Supplement (N=15) | Canola Oil Placebo (N=16)
Gastrointestinal Symptoms (Gastrointestinal disorders) | 10 | 11
Ear Nose Throat Symptoms (Ear and labyrinth disorders) | 6 | 9
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Skin and Limb Symptoms (Skin and subcutaneous tissue disorders) | 4 | 1
Behavioral Symptoms (Psychiatric disorders) | 3 | 3
Cold/Fever (Infections and infestations) | 2 | 5 — Multi-symptom illnesses reported by caregivers which typically included more than 1 body system and/or fever

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No